CLINICAL TRIAL: NCT01608854
Title: Prospective, Randomized Study of the Utilization of Antibiotics and Drains in Spinal Surgery
Brief Title: Comparison of Antibiotic Protocols in Spine Patients With Postoperative Drains
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: NYUHJD08139
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Surgical Wound Infection; Spinal Deformity; Spinal Degeneration
Keywords: surgical site infection; spinal surgery; prophylactic antibiotics; postoperative spinal drains
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 24 Hour Antibiotics: Patients were randomized to receive 24 hours of postoperative antibiotics following spine surgery
- Duration Antibiotics: Patients were randomized to receive antibiotics for the duration of time a spinal drain was in place following spinal surgery
  Interventions: Other: Antibiotic Protocol

INTERVENTIONS:
Other: Antibiotic Protocol — Patients were given postoperative antibiotics according to their randomization; antibiotic type and dosage were determined by the attending physician.
  Groups: Duration Antibiotics

SUMMARY:
In spine surgery, postoperative spinal drains are often utilized to prevent fluid buildup around the spinal cord. The purpose of this study is to determine whether postoperative antibiotic treatment continued for the duration of time a drain is in place results in a lower infection rate than antibiotics given for only 24 hours postoperatively.

DETAILED DESCRIPTION:
Patients likely to receive postoperative spinal drains were enrolled and randomized preoperatively to receive one of two postoperative antibiotic treatments, either for 24 hours after surgery or for the duration of time the spinal drain was in place. If patients did not receive at least one spinal drain during surgery, they were excluded from the infection analysis and received the institutional standard of 24 hours of postoperative antibiotics. Patients that did receive drains were treated according to their randomization and followed for a minimum of one year for the incidence of surgical site infection. The diagnosis of surgical site infection was determined using the definition provided for the Center for Disease Control (CDC). All patients that developed surgical site infections were treated as appropriate by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled to undergo spine surgery with likely drain placement (3 or more vertebral levels, dependent upon attending surgeon)
* Must be over the age of 18
* Must consent to randomized postoperative antibiotic treatment

Exclusion Criteria:

* Does not receive a drain at the time of surgery
* Surgery is cancelled
* Infection is present at the time of initial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical spine patients of a single urban institution from 2008-2011
Sampling Method: Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Infection | for one year after surgery
  Patients were contacted and their medical records were reviewed for a minimum of one year after surgery in order to determine the incidence of postoperative infection. The Center for Disease Control's definition of surgical site infection was applied in determining infection rates.

CONTACTS AND LOCATIONS:
Overall Officials: Baron S Lonner, MD, Principal Investigator — NYU Hospital for Joint Diseases
Locations (1):
- NYU Hospital for Joint Diseases, New York, New York, United States

REFERENCES:
- [Background] Brown MD, Brookfield KF. A randomized study of closed wound suction drainage for extensive lumbar spine surgery. Spine (Phila Pa 1976). 2004 May 15;29(10):1066-8. doi: 10.1097/00007632-200405150-00003. PMID 15131430
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Background] Drinkwater CJ, Neil MJ. Optimal timing of wound drain removal following total joint arthroplasty. J Arthroplasty. 1995 Apr;10(2):185-9. doi: 10.1016/s0883-5403(05)80125-1. PMID 7798099
- [Background] Fang A, Hu SS, Endres N, Bradford DS. Risk factors for infection after spinal surgery. Spine (Phila Pa 1976). 2005 Jun 15;30(12):1460-5. doi: 10.1097/01.brs.0000166532.58227.4f. PMID 15959380
- [Background] Fletcher N, Sofianos D, Berkes MB, Obremskey WT. Prevention of perioperative infection. J Bone Joint Surg Am. 2007 Jul;89(7):1605-18. doi: 10.2106/JBJS.F.00901. No abstract available. PMID 17606802
- [Background] Garcia S, Lozano ML, Gatell JM, Soriano E, Ramon R, Sanmiguel JG. Prophylaxis against infection. Single-dose cefonicid compared with multiple-dose cefamandole. J Bone Joint Surg Am. 1991 Aug;73(7):1044-8. PMID 1874767
- [Background] Glassman SD, Dimar JR, Puno RM, Johnson JR. Salvage of instrumental lumbar fusions complicated by surgical wound infection. Spine (Phila Pa 1976). 1996 Sep 15;21(18):2163-9. doi: 10.1097/00007632-199609150-00021. PMID 8893444
- [Background] Heydemann JS, Nelson CL. Short-term preventive antibiotics. Clin Orthop Relat Res. 1986 Apr;(205):184-7. PMID 3698375
- [Background] Ho C, Sucato DJ, Richards BS. Risk factors for the development of delayed infections following posterior spinal fusion and instrumentation in adolescent idiopathic scoliosis patients. Spine (Phila Pa 1976). 2007 Sep 15;32(20):2272-7. doi: 10.1097/BRS.0b013e31814b1c0b. PMID 17873822
- [Background] Lonstein J, Winter R, Moe J, Gaines D. Wound infection with Harrington instrumentation and spine fusion for scoliosis. Clin Orthop Relat Res. 1973 Oct;(96):222-33. No abstract available. PMID 4584242
- [Background] Massie JB, Heller JG, Abitbol JJ, McPherson D, Garfin SR. Postoperative posterior spinal wound infections. Clin Orthop Relat Res. 1992 Nov;(284):99-108. PMID 1395319
- [Background] Mauerhan DR, Nelson CL, Smith DL, Fitzgerald RH Jr, Slama TG, Petty RW, Jones RE, Evans RP. Prophylaxis against infection in total joint arthroplasty. One day of cefuroxime compared with three days of cefazolin. J Bone Joint Surg Am. 1994 Jan;76(1):39-45. doi: 10.2106/00004623-199401000-00006. PMID 8288664
- [Background] Nelson CL, Green TG, Porter RA, Warren RD. One day versus seven days of preventive antibiotic therapy in orthopedic surgery. Clin Orthop Relat Res. 1983 Jun;(176):258-63. PMID 6851335
- [Background] Parker MJ, Livingstone V, Clifton R, McKee A. Closed suction surgical wound drainage after orthopaedic surgery. Cochrane Database Syst Rev. 2007 Jul 18;2007(3):CD001825. doi: 10.1002/14651858.CD001825.pub2. PMID 17636687
- [Background] Parker MJ, Roberts CP, Hay D. Closed suction drainage for hip and knee arthroplasty. A meta-analysis. J Bone Joint Surg Am. 2004 Jun;86(6):1146-52. doi: 10.2106/00004623-200406000-00005. PMID 15173286
- [Background] Payne DH, Fischgrund JS, Herkowitz HN, Barry RL, Kurz LT, Montgomery DM. Efficacy of closed wound suction drainage after single-level lumbar laminectomy. J Spinal Disord. 1996 Oct;9(5):401-3. PMID 8938608
- [Background] Pollard JP, Hughes SP, Scott JE, Evans MJ, Benson MK. Antibiotic prophylaxis in total hip replacement. Br Med J. 1979 Mar 17;1(6165):707-9. doi: 10.1136/bmj.1.6165.707. PMID 373841
- [Background] Rello J, Sa-Borges M, Correa H, Leal SR, Baraibar J. Variations in etiology of ventilator-associated pneumonia across four treatment sites: implications for antimicrobial prescribing practices. Am J Respir Crit Care Med. 1999 Aug;160(2):608-13. doi: 10.1164/ajrccm.160.2.9812034. PMID 10430736
- [Background] Sankar B, Ray P, Rai J. Suction drain tip culture in orthopaedic surgery: a prospective study of 214 clean operations. Int Orthop. 2004 Oct;28(5):311-4. doi: 10.1007/s00264-004-0561-2. Epub 2004 Aug 14. PMID 15316674
- [Background] Sculco TP. The economic impact of infected joint arthroplasty. Orthopedics. 1995 Sep;18(9):871-3. No abstract available. PMID 8570494
- [Background] Thalgott JS, Cotler HB, Sasso RC, LaRocca H, Gardner V. Postoperative infections in spinal implants. Classification and analysis--a multicenter study. Spine (Phila Pa 1976). 1991 Aug;16(8):981-4. doi: 10.1097/00007632-199108000-00020. PMID 1948385
- [Background] Viola RW, King HA, Adler SM, Wilson CB. Delayed infection after elective spinal instrumentation and fusion. A retrospective analysis of eight cases. Spine (Phila Pa 1976). 1997 Oct 15;22(20):2444-50; discussion 2450-1. doi: 10.1097/00007632-199710150-00023. PMID 9355228
- [Background] Weinstein MA, McCabe JP, Cammisa FP Jr. Postoperative spinal wound infection: a review of 2,391 consecutive index procedures. J Spinal Disord. 2000 Oct;13(5):422-6. doi: 10.1097/00002517-200010000-00009. PMID 11052352
- [Background] Williams DN, Gustilo RB. The use of preventive antibiotics in orthopaedic surgery. Clin Orthop Relat Res. 1984 Nov;(190):83-8. PMID 6386263
- [Background] Wimmer C, Gluch H, Franzreb M, Ogon M. Predisposing factors for infection in spine surgery: a survey of 850 spinal procedures. J Spinal Disord. 1998 Apr;11(2):124-8. PMID 9588468